CLINICAL TRIAL: NCT02610023
Title: Comparative Assessment of Food Frequency Questionnaires
Brief Title: Food Frequency Questionnaires in Estimating Food Nutrient Intake in Healthy Young Adults
Status: Active, not recruiting | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Steven Clinton, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU 14222; NCI-2015-00069 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Healthy Subject
MeSH Terms: interventions — Spectrum Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observational (Willett FFQ, Fred Hutchinson FFQ, CCAT): After consenting to participate in this study, participants will visit the Clinical Research Center (CRC) on 3 occasions. One of the three FFQ's will be completed at each visit and there will be 4 to 6 weeks between visits. Participants will also complete a blood draw and assessment of skin carotenoids at this CRC visit. Prior to each visit, participants will complete a 3-day diet record, a daily sun exposure diary, and a 3-day activity record.
  Interventions: Other: Questionnaire Administration; Other: Laboratory Biomarker Analysis; Device: Spectroscopy

INTERVENTIONS:
Other: Questionnaire Administration — Complete the Willett FFQ, the Fred Hutchinson FFQ, and the CCAT
Other: Laboratory Biomarker Analysis — Correlative studies
Device: Spectroscopy — Undergo resonance Raman spectroscopy

SUMMARY:
Fruits and vegetables are an important source of many different phytochemicals that may affect health and accurate dietary assessement tools to quantitate dietary intake are essential. This study will evaluate the correlation of dietary carotenoid intake estimated from two common and one novel food frequency questionnaire (FFQ) with estimated carotenoid intake from 3 day diet records as well as measured blood and skin concentrations of carotenoids. This study will be conducted in healthy adults. These tools may be effective in estimating the level of these compounds in an average diet.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To examine the relationship between estimated intakes of dietary carotenoids using three different FFQ's and comparing them with estimated carotenoid intake from 3 day diet records and blood and skin measurements.

OUTLINE:

Participants complete the Willett FFQ, the Fred Hutchinson FFQ, and the newly developed Clinton Carotenoid Assessment Tool (CCAT), in random order over a 3 to 4-month period of time with 4-6 weeks between each visit. Prior to each visit, participants also complete a 3-day diet record, a daily sun exposure diary, and a 3-day activity record. Blood samples are collected for plasma carotenoid assessment and and skin carotenoid content is assessed using a resonance Raman spectroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Be literate and able to understand English
* Have a body mass index (BMI) between 18.5 and 30 kg/m^2; this represents the lowest end of the healthy BMI range and the upper limit of the overweight BMI range for our target age range
* Be a non-smoker (defined as adults who have never smoked or who have not had a cigarette in the past ten years)
* Not currently be taking any vitamins, minerals, or dietary supplements (or agree to discontinue use for the duration of the study) and agree to consume a standardized daily multivitamin for the remainder of the study (CVS One Daily)
* Voluntarily agree to participate and sign an informed consent document
* Agree to three separate blood draws
* Agree to three separate spectroscopy scans to assess skin carotenoid levels
* Agree to complete three separate 3-day diet records, three separate 3-day activity records, and one habitual physical activity questionnaire

Exclusion Criteria:

* Have an active metabolic or digestive illness, including malabsorptive disorders, renal insufficiency, hepatic insufficiency, hyper- or hypothyroidism, cachexia, morbid obesity, or short bowel syndrome
* Have an active or a recent history of any condition that causes altered immunity, such as chronic inflammatory disease, autoimmune disorders, cancer, anemia, and blood dyscrasias
* Are heavy alcohol consumers (defined as an average consumption of greater than 2 drinks/day)

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be recruited from the Ohio State University Campus, Wexner Medical Center Hospitals, and surrounding greater Columbus area.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
FFQ estimated carotenoid intake | Up to 3 months
  The relationship between the carotenoid values from the FFQ, both the unadjusted and the energy-adjusted estimates, and averages of the 3-day diet records will be estimated using the Pearson correlation coefficients. Statistical analysis will be conducted using Stata version 11.
Levels of carotenoids in plasma | Up to 3 months
  Pearson correlations will be used to compare plasma levels of individual carotenoids with their respective dietary intake after adjustment for total energy, plasma cholesterol, plasma triglycerides, and BMI. Statistical analysis will be conducted using Stata version 11.
CCAT ability to estimate carotenoid intake | Up to 3 months
  CCAT carotenoid intake will be correlated with blood carotenoid profiles. Statistical analysis will be conducted using Stata version 11.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Clinton, MD, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio, United States